CLINICAL TRIAL: NCT05858255
Title: Hjernegym - Effects of Exergaming in Psychosis: a Clinical Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Tom Langerud Holmen, Clinical Psychologist PhD, Sykehuset i Vestfold HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SykehusetIV
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Psychosis; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Exergaming; Exercise

STUDY DESIGN:
Intervention Model Description: Clinical intervention study
Masking Description: No masking is planned. A secondary aim of the study is to indicate the feasibility of the intervention in a daily clinical setting, with a minimum of additional assessments and involved personnel as compared to treatment as usual. Hence, the intervention will be conducted by designated personnel in line with all other treatment activities in the clinic, and (regular and additional) assessments will, for study purposes, be conducted by the PI instead of the participant's designated clinical team. Assessments and intervention sessions will however be conducted in close collaboration with the participants' designated clinical teams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergaming (Experimental): A 12-weeks, twice a week exergaming program, consisting of a combined high-intensity interval training and flash-reflex pods gaming condition, each session lasting 45 minutes, conducted one-on-one with a designated personal trainer (experienced and authorized health personnel with additional competence in exercise/sports and/or physical therapy).
  Interventions: Behavioral: Exergaming

INTERVENTIONS:
Behavioral: Exergaming — Please see Arms description.
  Other Names: Physical exercise

SUMMARY:
The goal of this clinical intervention study is to investigate the effects of exergaming on cognition and other clinical symptoms in outpatient individuals with schizophrenia.

The main questions it aims to answer are: Will an exergaming intervention contribute to improved cognition and reduced clinical symptoms, as well as enhanced physical health/self-efficacy/quality of life, in individuals with schizophrenia? Will the gaming component strengthen motivation for a physically more intensive component, so that attendance will be at least as high as in comparable exercise studies despite the current study being implemented in a resource-limited, regular clinical outpatient setting? Participants will be asked to engage in two 45 minutes exergaming sessions with a designated personal trainer for 12 weeks. Results pre- and post intervention will be compared, and comparisons will also be made with a former randomized controlled trial conducted at the same site, in which the currently combined activities were investigated separately (high-intensity interval training and low-intensity video gaming), both yielding positive but different effects.

DETAILED DESCRIPTION:
Cognitive impairment is a core clinical feature in schizophrenia, central to the affected individuals' daily functioning. Regular treatment components such as medication or psychotherapy provide no effective remediation for this. However, research has shown that both high-intensity interval training (HIIT) and active video gaming (AVG) may have beneficial effects on cognitive functioning, and also other clinical symptoms, for individuals with schizophrenia. Moreover, the two activity types yield partly overlapping, partly differentiated effects on these outcome measures: While the former may improve cognitive functions through enhanced cardio-respiratory fitness, the latter may facilitate synapto-genesis through learning of new motor- and coordination patterns. Furthermore, HIIT may counter depressive symptoms while AVG may strengthen motivation for regular activity. Results consistent with this was found in the randomized controlled trial "Effects of Physical Activity on Psychosis" (EPHAPS) previously conducted at the same site as the currently planned study (DPS Vestfold, the psychosis outpatient clinic, 2014 - 2017). Hence, the two activity types combined - "exergaming" - may have complementary positive effects on cognition and other clinical symptoms, as well as physical health, while also facilitating the participants' motivation for regular attendance. This assumption is supported by the few existing studies on exergaming interventions for individuals with schizophrenia. However, research into this area is yet scarce. Based on the existing evidence for the two activity types both separately and combined, exergaming alternatives are already being tested out in the clinic at DPS Vestfold. To meet the need for more research in this area, the investigators plan to include 48 participants in an exergaming clinical intervention study. By implementing such a study in a regular clinical setting and with the least amount of additional resources possible, the investigators also seek to demonstrate the intervention's feasibility for individuals with schizophrenia. Upon supported research hypotheses, the intervention could easily be adapted to similar clinical settings and included as a standard care-component.

ELIGIBILITY:
Inclusion Criteria:

* Having consent capability
* Understanding and speaking Scandinavian language
* Fulfilling the International Classification of Diseases Tenth Revision (ICD 10) criteria for schizophrenia spectrum disorder (schizophrenia, schizoaffective disorder and schizophreniform disorder)

Exclusion Criteria:

* Diagnosis of intellectual disability
* Diagnosis of neurological disorder
* History of severe head trauma
* Pregnancy
* Chest pain during exercise
* Unstable angina pectoris
* Malignant hypertension
* Uncontrollable arrhythmia
* Recent myocardial infarction
* Acute infection with lymphadenopathy
* Other specified medical condition incompatible with participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved cognition as measured by increased scores on the MCCB test battery. | Baseline and 12 weeks.
  Cognitive improvement as measured by increased scores on the Matrics Consensus Cognitive Battery (MCCB) (except for the omitted MSCEIT social cognition test); changes in scores of each of the nine subtests as well as the total (neurocognitive composite-) score will be evaluated.
Sustained motivation for the intervention activity (exergaming) as measured by high attendance/adherence to protocol and low levels of drop-out/withdrawal, respectively. | 12 weeks.
  High attendance/adherence to protocol and low dropout/withdrawal as evaluated against a comparable exercise study conducted at the same site (dropout/withdrawal rate equal to or below 15%), with the current study being implemented in a resource-limited, regular clinical setting. These may serve as indicators of the gaming component's motivating potential for the more physically demanding elements in the intervention activity, and also the feasibility and economical viability of the activity as a regular treatment component for individuals with schizophrenia spectrum disorders.

SECONDARY OUTCOMES:
Reduced depressive- and other symptoms as measured by the PANSS interview. | Baseline and 12 weeks.
  Reduction in symptom scores on the Positive and Negative Syndrome Scale; changes in scores on each of the five symptom domains of the widely used PANSS five factor consensus model suggested by Wallwork et al., as well as the total PANSS score, will be evaluated.
Reduced levels of self-disorders as measured by the EASE interview. | Baseline and 12 weeks.
  Reduction in levels of self-disorders as measured by reduced total score on the Examination of Anomalous Self-Experience interview (contingent on proper certification of the assessor/PI, for the use of the interview).
Improved oxygen consumption as measured by a VO2peak-test. | Baseline and 12 weeks.
  Increased oxygen consumption as indicated by higher scores on a VO2peak-test (a maximum exercise test on a treadmill utilizing a modified Balke protocol): Gas exchange sampled continuously (mixing chamber every 30 s); two-ways breathing valve connected to a gas analyser measuring oxygen - carbon dioxide content.

OTHER OUTCOMES:
Improved self-efficacy as measured by the GSE. | Baseline and 12 weeks.
  Increased levels of self-efficacy as indicated by higher scores on the Generally Perceived Self-Efficacy Scale.
Improved quality of life as measured by the SF-12 questionnaire. | Baseline and 12 weeks.
  Increased experienced quality of life as indicated by higher scores on the RAND 12 Short Form Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Langerud Holmen, PhD, Principal Investigator — Sykehuset i Vestfold HF
Locations (1):
- DPS Vestfold, Vestfold Sykehus HF, Tønsberg, Vestfold, Norway

IPD SHARING:
Plan to Share IPD: No
Due to restrictions on sensitive health data, the investigators are not able to openly share these data with other researchers outside the organization.